CLINICAL TRIAL: NCT05338138
Title: Point of Care Ultrasonography Versus Standard Blind Technique for Central Venous Catheter Insertion in Emergency Hospital
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ahmed Beniamen Mohamed Hussien, lecturer of anethesia and icu faculty of medicine zagazig university, Zagazig University
Other Study IDs: ZU-IRB#:6827/30-3-2021
Record Dates: First submitted 2022-04-08; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Central Venous Catheter Placement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- the standard blind technique for Central venous catheter insertion into the internal jugular vein.: using the blind experience based technique without imaging guidance
- ultrasound guided technique for Central venous catheter insertion into the internal jugular vein.: using real time ulrasound guidance
  Interventions: Device: ultrasound guided central venous catheter insertion

INTERVENTIONS:
Device: ultrasound guided central venous catheter insertion — Prospective comparative randomized controlled clinical study.
  Groups: ultrasound guided technique for Central venous catheter insertion into the internal jugular vein.

SUMMARY:
A lot of complications occur during central venous catheter insertion in intensive care units all over the world most commonly pneumothorax, misplacement and infection. So in this study we will assess the effect of using ultrasonography guidance for CVC insertion to reduce incidence of complications and to confirm placement compared to standard blind technique.

DETAILED DESCRIPTION:
Central venous catheter (CVC) - also called central venous access, central venous line, or central line - is a thin catheter that is inserted through one of the large veins in the neck area into the venous system. It ends in one of the venae cavae just before entering the right atrium.

CVC is a procedure frequently required in critical care units. Indications include patients with multiple, incompatible intravenous (IV) medications with limited peripheral access, or who are being treated with vasoactive or phlebosclerotic agents which may not be suitably cared for with a peripheral IV alone. Some central lines are also placed for temporary or permanent hemodialysis access; these dialysis catheters are significantly larger than traditional double, triple, or quadruple lumen catheters placed in the emergency department or intensive care unit setting.

Central lines are placed today via the Seldinger technique, in which the chosen vein is cannulated with a needle, a guidewire is inserted to maintain a tract through the skin into the vein, and the catheter is then inserted over the wire into the vein before the wire is removed. When this procedure was performed blindly it was called the standard technique, while if it was done with ultrasound guidance it is called ultrasound guided technique.

Patients were selected from emergency hospital at zagazig university hospitals who needed CVC insertion as an important part of management plan

All Cases underwent:

1. Patient Examination: regarding written consent from patients or relatives when possible, site of planned insertion, explanation to the patient if conscious and cooperative and checking platelet count and INR if available (not necessary in emergency situation)
2. Randomization: A computer-generated randomization table allocated the patients into 2 equal groups.
3. Preparation: Once the site was chosen, a topical antiseptic such as chlorhexidine or betadine was applied circularly to the skin in ever-enlarging circles. Once applied, the antiseptic was allowed to dry to maximize the decrease in skin surface bacterial cell count. After securing the line in vivo, it was also common practice to flush the central line with sterile saline to prevent clotting within the catheter, as well as to confirm the functionality of all ports. This step was performed both prior to insertion and after insertion of the catheter.
4. Personnel: When possible, having an assistant present during the procedure was helpful.
5. Equipment for CVC insertion:

   * Central line insertion kit, which is usually manufacturer-specific should contain the all the equipment for the central line and Seldinger technique, including a central venous catheter, guidewire, syringe, an introducer needle, a scalpel, a silk suture (on a Keith or curved needle) and a skin dilator
   * Sterile gloves and gown
   * Hat and mask
   * Drape or sterile towels to create a sterile barrier (to protect equipment and materials from becoming contaminated)
   * Antiseptic agent for skin preparation
   * Proper caps for each lumen port
   * Dressing to cover the insertion site
   * Local anesthetic (1% to 2% lidocaine)
   * If an ultrasound-guided technique was used, a sterile probe cover was used.
6. Technique:

In group A: the insertion site was anesthetized by injecting local anesthetic sufficient to create a wheal under the skin. then the needle was advanced towards the venous target, aspirating then injecting anesthetic into the subcutaneous tissue. Once the area is anesthetized, the introducer needle was introduced into the skin, and advanced toward the vein being cannulated, all the while aspirating with steady pressure. then continued as seldinger maneuver In group B: the ultrasound machine was employed using the linear probe, the probe was covered by a sterile cover, and then localization of internal jugular vein (IJV) was done. The IJV was adjusted to be at the center of the ultrasound monitor view then slight compression on IJV was done to ensure its patency and collapsibility and to differentiate IJV from carotid artery that should be visualized beside or behind the IJV as a pulsating non collapsible vessel that colors red on Doppler while the IJV colors blue on Doppler. then the next steps were continued as the standard blind technique. Immediately after CVC placement, a saline flush consisting of 10 mL of normal saline was injected into the distal hub of the CVC by the interventionist while focused echocardiography was conducted by a second resident. The time required for the procedure was recorded. Appearance of an opacification of the right atrium (RASS) was judged as "immediate" (less than two seconds after injection), "delayed" (appearing more than two seconds after injection) or "absent". Echocardiography was immediately evaluated by the resident placing the catheter and the result ("delayed", "immediate" or "absent" flush) recorded by one investigator (EM). The examination was repeated up to three times and catheter position corrected during placement when the saline flush test was indicative of a problem. Overall, a positive RASS (negative screening test for misplacement) translated into a correctly positioned catheter, whereas a delayed or absent flush (negative RASS or positive screening test) implied a potentially misplaced catheter (Korsten et al., 2018).

After CVC insertion was finished, chest ultrasonography was done by the intensivist to exclude presence of pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

1. Patient acceptance (if conscious)
2. Aged >18years.
3. Gender: both.

5. Patients admitted to emergency hospital units, at emergency room (ER), operation theater (OT) or emergency intensive care unit (ICU)

Exclusion Criteria:

1. Patient refusal
2. Coagulopathy: INR>1.5 or platelet count<500000/cc
3. Skin infection at site of insertion
4. Physician not well trained on utilization of ultrasound machine or even not familiar with it.
5. History of surgical manipulation or trauma at the insertion site
6. Trauma to other structures (e.g. cervical spine collar is a soft contraindication to an IJ central venous catheter (CVC) placement, a pelvic binder is a contraindication to a femoral CVC placement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from emergency hospital at zagazig university hospitals who needed CVC insertion as an important part of management plan.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
the incidence of complications in ultrasound guided central venous catheter insertion | 6 months from october 2021 to april 2022
  the incidence of complications in ultrasound guided central venous catheter insertion is expected to be lower than the standard blind technique

CONTACTS AND LOCATIONS:
Overall Officials: ahmed B mohamed, MD, Principal Investigator — Zagazig University
Locations (1):
- ZagazigU, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
protocol only